CLINICAL TRIAL: NCT01556568
Title: An Open Label Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MEK162 in Noonan Syndrome Hypertrophic Cardiomyopathy
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MEK162 in Noonan Syndrome Hypertrophic Cardiomyopathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to scientific and business considerations.
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162Y2201; 2011-003392-10 (EudraCT Number)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Cardiomegaly
Keywords: Noonan Syndrome, hypertrophic cardiomyopathy.
MeSH Terms: conditions — Cardiomegaly; Noonan Syndrome; Cardiomyopathy, Hypertrophic | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEK162 (Experimental): Patients will be treated with MEK162 only and will be uptitrated or down titrated based on safety and tolerability observed.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162

SUMMARY:
The purpose of the study is to determine whether the ability of MEK162 to antagonize MEK activation in NS HCM patients, who usually have upstream mutations in the Ras-Raf-Mek-Erk pathway that lead to MEK activation, would be beneficial over a 6 month treatment period in hypertrophy regression.

DETAILED DESCRIPTION:
This study is designed as a proof of concept of MEK162 in NS HCM patients. The purpose of the present study is to determine whether the ability of MEK162 to antagonize MEK activation in NS HCM patients, who usually have upstream mutations in the Ras-Raf-Mek-Erk pathway that lead to MEK activation, would be beneficial over a 6 month treatment period by causing hypertrophy regression. Such regression might result in cardiovascular clinical benefits with longer term treatment.

The information gained from this study will be three fold:

1. the safety/tolerability of treatment with MEK162 over 6 month in the NS HCM patient population
2. the pharmacokinetics and pharmacodynamics of MEK162 in the target patient population
3. proof of the therapeutic concept that MEK inhibition will reduce cardiac hypertrophy in the target NS HCM patient population

ELIGIBILITY:
Inclusion:

* Male and female Noonan syndrome patients with confirmed cardiac hypertrophy, age 18 to 65 years of age included, and in general good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Cardiac hypertrophy is defined by left ventricular wall thickness greater than or equal to 12 mm by echocardiography or MRI, or the change in wall thickness is accompanied by an associated increase in left ventricular mass which is defined by echo or MRI as greater than 134 g/m2 and 110 g/m2 in men and women, respectively.
* Subjects must weigh at least 45 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 34 kg/m2.

Exclusion criteria:

* Primary Long QT syndrome or a history of significant ECG abnormalities judged by the investigators to be inappropriate for participation in the current study.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Sexually active males must use a condom during intercourse while taking the drug during treatment, for 5 half lives after stopping treatment and should not father a child in this period.
* Use of any prescription drugs other than beta-blockers, diuretics, CCB, amiodarone, disopyramide, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing. If needed, (i.e. an incidental and limited need) paracetamol or acetaminophen is acceptable, but must be documented in the Concomitant medications/Significant non-drug therapies page of the eCRF.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Left ventricular mass (LVM) | Baseline to 3 months and 6 months
  Change in LVM after 3 months and 6 months of treatment using magnetic resonance imaging.

SECONDARY OUTCOMES:
Change from baseline in Cardiac energetics state at 3 months and 6 months | Baseline to 3 months and 6 months
  Energetic state represented by phosphocreatine (PCr)/adenosine triphosphate (ATP) ratio using magnetic resonance spectroscopy.
Number of patients with adverse events, serious adverse events and death | 6 months
  Abnormalities in Vital signs, ECG evaluations, clinical laboratory evaluations, will be collected.
Pharmacokinetics of MEK162 and metabolite (AR00426032): The trough plasma concentration (Ctrough) just prior to drug administration | Days 1, 8, 15, 28, 56, 84, 140 and 182
  pre-dose concentration of MEK162 and its metabolite (AR00426032) in plasma. All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Pharmacokinetics of MEK162 and metabolite (AR00426032): maximum drug exposure of MEK162 and its metabolite (AR00426032) in plasma | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Pharmacokinetics of MEK162 and metabolite (AR00426032): time to reach peak concentration (Tmax) in plasma | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Pharmacokinetics of MEK162 and metabolite (AR00426032): Area under the plasma concentration-time profile from time zero to 12 hours post dose (AUC0-12h) | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Pharmacokinetics of MEK162 and metabolite (AR00426032): Area under the plasma concentration-time profile from time zero to the last quantifiable sample (AUClast) | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Pharmacokinetics of MEK162 and metabolite (AR00426032): accumulation ratio (Racc) | Day 1 and Day 8
  Comparison of the drug exposures as AUCs and Cmax of MEK162 and its metabolite (AR00426032) in plasma after 8 days treatment in relation to the data from the first day (Day 8/Day 1)
Pharmacokinetics of MEK162: The degree of fluctuation of MEK162 and its metabolite (AR00426032) in plasma at steady state (on Day 8) | Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein. The dgree of fluctuation is calculated as (Cmax,ss - Cmin,ss)/Cav,ss at steady state.
Pharmacokinetics of MEK162: The ratio of Metabolite (AR00426032) to MEK162 in plasma on Days 1 and 8 | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Change from baseline in end systolic and end diastolic right and left vetricular volumes in 3 and 6 months | baseline to 3 and 6 months of treatment
  These parameters are derived from cine breath-hold magnetic resonance images acquired over the cardiac cycle.
Pharmacokinetics of MEK162 and metabolite (AR00426032):observed maximum plasma concentration (Cmax) following drug adminstration | Day 1 and Day 8
  All blood samples will be taken by either direct venipuncture or an indwelling cannula inserted in a forearm vein.
Change from baseline in stroke volume and stroke output during 3 and 6 months | baseline to 3 and 6 months of treatment
  These parameters are derived from cine breath-hold magnetic resonance images acquired over the cardiac cycle.
Ejection fraction | baseline, 3 and 6 months of treatment
  This parameter is derived from cine breath-hold magnetic resonance images acquired over the cardiac cycle.
Cardiac index | baseline, 3 and 6 months of treatment
  This parameters is derived from cine breath-hold magnetic resonance images acquired over the cardiac cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigative Site, Boston, Massachusetts, United States
- Pfizer Investigative Site, London, United Kingdom